CLINICAL TRIAL: NCT07310654
Title: Effects of a 16-week Moderate-to-Vigorous Physical Activity Program on Physical Fitness and Gut Microbiota in Children: A Randomized Controlled Trial
Brief Title: Physical Activity and Gut Microbiota in Children (PA-Microbiome Kids)
Acronym: PA-Microbiome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aiyoudong Children and Youth Sports Health Research Institute (Other)
Responsible Party: Principal Investigator, Pan Xiang, Researcher, Aiyoudong Children and Youth Sports Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PA-Microbiome-Kids-2025; 2244 (Other Grant/Funding Number: China Institute of Sport Science)
Record Dates: First submitted 2025-12-03; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: Physical Activity; Gut Microbiota; Microbiome; Physical Fitness; Children; Health Promotion
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and intervention instructors are not blinded to group assignment. Outcome assessors (for physical fitness tests) and laboratory/bioinformatics personnel (for microbiota analysis) will be blinded to the allocation. The database will use codes (e.g., Group A/B) until primary analysis is complete.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MVPA Program (Experimental): Participants will engage in a 16-week structured moderate-to-vigorous physical activity (MVPA) program, 3 times per week, for 45-60 minutes per session. Sessions include warm-up, aerobic games, bodyweight strength circuits, and cool-down, supervised by trained instructors.
  Interventions: Behavioral: 16-week Structured MVPA Program
- : Attention Control + Waitlist (Active Comparator): Participants will engage in time-matched sedentary activities, such as reading, science experiments, or crafts, 3 times per week. They are instructed to maintain their usual physical activity levels. After the 16-week trial period, they will be offered a similar MVPA program.
  Interventions: Behavioral: Attention Control Sedentary Activities

INTERVENTIONS:
Behavioral: 16-week Structured MVPA Program — A 16-week structured moderate-to-vigorous physical activity program.
  Arms: MVPA Program
Behavioral: Attention Control Sedentary Activities — Time-matched sedentary activities such as reading, science experiments, or crafts.
  Arms: : Attention Control + Waitlist

SUMMARY:
This study evaluates the effect of a 16-week moderate-to-vigorous physical activity (MVPA) program on physical fitness and gut microbiota in healthy school-aged children. Participants will be randomly assigned to either an MVPA intervention group or an attention-control group. The primary outcome is the change in a composite physical fitness score. Secondary outcomes include changes in gut microbiota diversity and composition.

DETAILED DESCRIPTION:
This is a two-arm, parallel-group, randomized controlled trial with 1:1 allocation. Healthy children aged 7-10 years will be recruited. The intervention group will receive a 16-week structured MVPA program (3 sessions/week, 45-60 min/session). The control group will receive attention-matched sedentary activities (e.g., reading, crafts) and will be offered the MVPA program after the trial (waitlist). Blinding will be applied to outcome assessors and laboratory/bioinformatics analysts. The primary analysis will follow the intention-to-treat (ITT) principle. The study aims to determine if the MVPA intervention improves physical fitness and modulates the gut microbiota, and to explore baseline microbiota features as potential modifiers of the intervention response.

ELIGIBILITY:
Inclusion Criteria:

* Participants from a previous cross-sectional study cohort conducted in August 2024, at which time they were 6-9 years old.
* Able to complete the 16-week follow-up.
* Guardian provides written informed consent, and the child provides assent.
* Medically cleared by a physician or school nurse to participate in moderate-intensity physical activity (no contraindications).
* No antibiotic use in the 4 weeks prior to baseline.
* No fever or acute gastroenteritis in the 2 weeks prior to baseline.
* Able to provide stool samples as required.

Exclusion Criteria:

* Diagnosed with cardiopulmonary diseases, epilepsy, severe asthma, severe musculoskeletal disorders, or congenital heart disease.

  * Recent acute exacerbation of chronic gastrointestinal diseases.
  * Planning to follow a special diet (e.g., ketogenic, vegetarian) or requiring long-term prescription of antibiotics/probiotics.
  * Planning to be absent for >20% of the intervention period due to travel or other commitments.
  * Enrolled in other high-intensity sports training programs that cannot be cancelled.
  * Developmental or behavioral issues that would impede cooperation, as assessed by teachers and parents.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 113 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Composite Physical Fitness Z-score | Baseline and 16 weeks
  Change from Baseline to 16 weeks in a composite physical fitness z-score. The score is calculated based on the age-appropriate items and weighting from the "National Student Physical Health Standard (2014 Revision)". The scale is a standardized z-score with a mean of 0 and a standard deviation of 1, based on a reference population. There are no theoretical upper or lower limits, but values typically range from -3 to +3. A higher score indicates better overall physical fitness.

SECONDARY OUTCOMES:
Change in Gut Microbiota Alpha Diversity | Baseline and 16 weeks
  Change from Baseline to 16 weeks in alpha diversity indices (Shannon and Chao1) of the gut microbiota, assessed via 16S rRNA gene sequencing. The Shannon index has a minimum value of 0, with no theoretical maximum. The Chao1 index estimates species richness with a minimum equal to the number of observed species, and also has no theoretical maximum. For both indices, higher values indicate greater diversity and are generally considered to reflect a healthier gut microbiome.
Difference in Gut Microbiota Beta Diversity | Baseline and 16 weeks
  Difference in gut microbiota community structure (beta diversity) between the MVPA and control groups. This will be assessed using a Permutational Multivariate Analysis of Variance (PERMANOVA) on Bray-Curtis and UniFrac distance matrices. The outcome will be reported as an R-squared value, representing the percentage of variance in community structure explained by group assignment, and a p-value. A larger R-squared value and a smaller p-value would indicate a more significant difference between the groups.
Change in Body Mass Index (BMI) Z-score | Baseline and 16 weeks
  Change from Baseline to 16 weeks in age- and sex-specific BMI z-score. This is a standardized score with a mean of 0, based on a reference population, and has no theoretical upper or lower limits. A higher score indicates a higher BMI relative to peers. In the context of this study focusing on healthy weight, an increase in the z-score is generally considered a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Aiyoudong Children and Youth Sports Health Research Institute, Weifang, Shandong, China

IPD SHARING:
Plan to Share IPD: No